CLINICAL TRIAL: NCT03787888
Title: Frequency of Hyponatremia Caused by Polyethylene Glycol Solution When Used as a Bowel Cleansing Agent for Colonoscopy
Brief Title: Hyponatremia Due to Poly Ethylene Glycol (PEG)
Status: Completed | Type: Observational
Sponsor: Tazeen Rasheed (Other)
Responsible Party: Sponsor-Investigator, Tazeen Rasheed, Assistant Professor, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Other Study IDs: DUHS
Record Dates: First submitted 2018-12-15; First posted 2018-12-26 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2018-12

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colonoscopy is a useful tool used in modern medicine and it is increasingly being employed for both diagnostic and therapeutic purposes. (Polyethelene glycol)PEG is very often used for bowel preparation.There are some cases of hyponatremia reported due to the use of PEG. This study was designed to find frequency of sodium disorders after bowel cleansing by Polyethylene glycol solution for colonoscopies in Dr. Ruth K.M. Pfau, Civil Hospital Karachi.

DETAILED DESCRIPTION:
Colonoscopy is a useful tool used in modern medicine and it is increasingly being employed for both diagnostic and therapeutic purposes. PEG is very often used for bowel preparation. PEG solutions clean the bowel with less water and electrolyte shifts, primarily by causing mechanical effect of large-volume lavage 1. However, there are some cases of hyponatremia reported due to the use of PEG. Life-threatening fluid and electrolyte disturbances are more likely to occur in patients with risk factors, such as old age, use of SSRIs and thiazide diuretics, chronic kidney disease, congestive heart failure or with a history of electrolyte abnormalities 2.

Although sporadic case reports of hyponatremia and other electrolyte imbalances after bowel preparation have been reported, but well-designed studies are lacking on this subject. Literature search did not reveal any local studies on this subject. This study was designed to find frequency of sodium disorders after bowel cleansing by Polyethylene glycol solution for colonoscopies in Dr. Ruth K.M. Pfau, Civil Hospital Karachi.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender of age between 18-80 years undergoing colonoscopy.
2. Patients should have normal electrolytes before taking solution.
3. Patients should have given informed consent.
4. Patients should have taken solution adequately before procedure.

Exclusion Criteria:

1. Patients with chronic kidney disease
2. Patients on diuretics
3. Patients who are hyponatremic on first sample, i.e., before taking bowel cleansing agent.
4. Hypothyroidism

   -

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopy at OT complex Dr. K.M. Pfau, Civil Hospital Karachi.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of hyponatremia caused by polyethelene glycol. | 12 hours
  Frequency of hyponatremia caused by polyethelene glycol when used as a bowel cleansing agent for colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Haris Alvi, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Ruth KM Pauf Civil Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] ASGE Technology Committee; Mamula P, Adler DG, Conway JD, Diehl DL, Farraye FA, Kantsevoy SV, Kaul V, Kethu SR, Kwon RS, Rodriguez SA, Tierney WM. Colonoscopy preparation. Gastrointest Endosc. 2009 Jun;69(7):1201-9. doi: 10.1016/j.gie.2009.01.035. No abstract available. PMID 19481646
- [Background] Samad N, Fraser I. Severe symptomatic hyponatremia associated with the use of polyethylene glycol-based bowel preparation. Endocrinol Diabetes Metab Case Rep. 2017 Feb 23;2017:16-0119. doi: 10.1530/EDM-16-0119. eCollection 2017. PMID 28458891